CLINICAL TRIAL: NCT06715059
Title: Effects of Tele-rehabilitation on Inter-Recti Distance, Postural Balance, Abdominal Endurance and Pelvic Floor Functions
Brief Title: Tele-rehabilitation in Women With Diastasis Recti Abdominis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assistant Professor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hdenizkulli
Record Dates: First submitted 2024-11-21; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Diastasis Recti; Diastasis Recti and Weakness of the Linea Alba
Keywords: inter-recti distance; postural control; pelvic floor dysfunction; body-self relation; abdominal endurance
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehab group (Experimental): The participants who performed exercise program via online platform.
  Interventions: Other: Tele-rehabilitation exercise program
- Home-based group (Experimental): The participants who performed exercise program in the home.
  Interventions: Other: Home-based exercise program

INTERVENTIONS:
Other: Tele-rehabilitation exercise program — A progressive core stability exercise program will be performed based on motor control principles via an online platform.
  Arms: Tele-rehab group
Other: Home-based exercise program — A core stability exercise program will be performed at home.
  Arms: Home-based group

SUMMARY:
The aim of this randomized controlled study is to determine the effect of motor-control based telerehabilitation exercise program on inter-recti distance, abdominal endurance, pelvic floor dysfunction, and body-image perception in women with diastasis recti abdominis.

Researchers will compare the effects of motor-control-based telerehabilitation exercise program and conventional exercise programs in women with DRA.

DETAILED DESCRIPTION:
Diastasis of recti abdominis (DRA) is defined as a separation of the two rectus abdominis muscles along the linea alba. Increased volume in the abdominal cavity, hormonal changes during pregnancy, neurodevelopmental differences, or abdominal wall laxity may caused. It is very common during pregnancy and may continue in the postnatal period. The loss of abdominal wall stability and weakened pelvic floor muscles may occur with DRA. The abdominal wall is one of the key point for body posture, trunk and pelvic stability. The core stability exercises, pelvic floor training and trunk muscle trainings are some of the exercise regimes options for management of DRA. However, in our best knowledge, there is no study in the literature that evaluates the effect of motor-control based telerehabilitation exercise program in women with DRA.

ELIGIBILITY:
Inclusion Criteria:

* Post- partum women (min 1 - max 5 years)

Exclusion Criteria:

* Having a neurological, orthopedical or any other condition which affect postural stability.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Inter-recti distance | baseline
  The subjects are assessed the inter-recti distance (IRD) in the supine position, knees bent and feet resting position on the table, the subjects is going to be asked to elevate the head and shoulders upwards until the inferior angles of the scapulae were just off the table.The subjects palpated the medial edges of RA muscles and IRD was measured using finger palpation in previously marked five-point: on the umbilicus, 5 cm, and 2 cm above and below the umbilicus
Inter-recti distance | after 8 weeks
  The subjects are assessed the inter-recti distance (IRD) in the supine position, knees bent and feet resting position on the table, the subjects is going to be asked to elevate the head and shoulders upwards until the inferior angles of the scapulae were just off the table.The subjects palpated the medial edges of RA muscles and IRD was measured using finger palpation in previously marked five-point: on the umbilicus, 5 cm, and 2 cm above and below the umbilicus

SECONDARY OUTCOMES:
Abdominal muscle endurance test | baseline
  The static abdominal flexion endurance test is also performed once in the same position as the IRD test. The subjects are asked to raise their head and shoulders upwards until the scapulae cleared the table and keep the position as long as possible. The time was recorded as the score of the test.
Abdominal muscle endurance test | After 8 weeks
  The static abdominal flexion endurance test is also performed once in the same position as the IRD test. The subjects are asked to raise their head and shoulders upwards until the scapulae cleared the table and keep the position as long as possible. The time was recorded as the score of the test.
Pelvic floor dysfunction | baseline
  Every subject will complete the Turkish version of the short-form of Pelvic Floor Distress Inventory (PFDI-20) which consists of three subscales: the Pelvic Organ Prolapse Distress Inventory short-form (POPDI6), the Urogenital Distress Inventory short-form (UDI-6), and the Colorectal-Anal Distress Inventory short-form (CRADI-8) to assess prolapse and pelvic pressure, urinary symptoms, and bowel symptoms, respectively
Pelvic floor dysfunction | After 8 weeks
  Every subject will complete the Turkish version of the short-form of Pelvic Floor Distress Inventory (PFDI-20) which consists of three subscales: the Pelvic Organ Prolapse Distress Inventory short-form (POPDI6), the Urogenital Distress Inventory short-form (UDI-6), and the Colorectal-Anal Distress Inventory short-form (CRADI-8) to assess prolapse and pelvic pressure, urinary symptoms, and bowel symptoms, respectively
Body-self relation | baseline
  Every subject will complete the Turkish version of Multi-Dimensional Body-Self Relations Questionnaire.
Body-self relation | After 8 weeks
  Every subject will complete the Turkish version of Multi-Dimensional Body-Self Relations Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal DENİZOĞLU KÜLLİ, Principal Investigator — İSTANBUL ATLAS ÜNİVERSİTESİ
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Atlas University, Istanbul, KAgıthane
  - Atlas University, Istanbul, Kağıthane